CLINICAL TRIAL: NCT01746511
Title: The Use of Glycerin Suppositories to Reduce Hyperbilirubinemia in Premature Infants Requiring Phototherapy
Brief Title: Glycerin Suppositories to Reduce Jaundice in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Carl D'Angio, Associate Professor of Pediatrics, Neonatology and Medical Humanities; Director, Neonatal Clinical Research; Director, Pediatric Clinical Research Office, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RSRB00040723
Record Dates: First submitted 2012-10-08; First posted 2012-12-11 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-11

CONDITIONS: Idiopathic Hyperbilirubinemia; Neonatal Hyperbilirubinemia; Prematurity
Keywords: glycerin suppositories; glycerin shaves; neonatal hyperbilirubinemia; idiopathic hyperbilirubinemia; jaundice; neonatal jaundice; prematurity
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Premature Birth; Jaundice; Jaundice, Neonatal | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glycerin Suppository (Active Comparator): Based on our institution's protocol, infant will receive a glycerin shave within one hour of initiation of phototherapy and then every eight hours while under phototherapy.
  Subjects will be block randomized (varying block sizes of 2 to 8). Babies in both groups will be fed according to NICU standard birth weight protocols. Stratified enrollment will occur with 2 separate groups:
  1. Infants who are NPO (< 20 mL/kg/day of fluids enterally at the time of therapy) vs.
  2. Those being enterally fed at least 20 mL/kg/day of total fluids at the time of therapy.
  Interventions: Procedure: Phototherapy; Drug: glycerin suppository
- No Glycerin Suppository (Experimental): Infants will receive no scheduled glycerin suppositories, while under phototherapy (unless otherwise directed by attending physician).
  Subjects will be block randomized (varying block sizes of 2 to 8). Babies in both groups will be fed according to NICU standard birth weight protocols. Stratified enrollment will occur with 2 separate groups:
  1. Infants who are NPO (< 20 mL/kg/day of fluids enterally at the time of therapy) vs.
  2. Those being enterally fed at least 20 mL/kg/day of total fluids at the time of therapy.
  Interventions: Procedure: Phototherapy

INTERVENTIONS:
Procedure: Phototherapy — Light therapy is used to treat cases of neonatal jaundice through the isomerization of the bilirubin and consequently transformation into compounds that the newborn can excrete via urine and stools.
  Other Names: Bili light
Drug: glycerin suppository — Promotes stooling through rectal stimulation and softening of stool. Given every 8 hours rectally. A pediatric glycerin suppository is 1.2 grams. All infants in this study arm will receive our standard dose of glycerin suppository which is 0.25 of the pediatric suppository or 0.3 grams.
  Other Names: glycerin shave
  Arms: Glycerin Suppository

SUMMARY:
The purpose of this study is to find out if giving glycerin suppositories will help decrease the length of time premature infants need phototherapy.

The investigators hypothesize that glycerin suppositories (initiated along with phototherapy) will have no effect on reducing duration of phototherapy in premature infants with jaundice.

DETAILED DESCRIPTION:
Neonatal jaundice is one of the most common clinical problems in the neonatal period (Maisels). Physiologic hyperbilirubinemia is usually benign and transient in nature. Bilirubin overproduction, delayed hepatic clearance, and increased enterohepatic circulation of bilirubin all contribute to neonatal jaundice (Bader). Previous studies have shown that delayed meconium evacuation might be an important contributing factor in the development and persistence of neonatal jaundice (Rosta and Porto). Once conjugated bilirubin is excreted from the liver to the small intestine, it is often deconjugated in the presence of alkaline media and beta-glucorinase enzymes which are present in abundance in premature infants. Once deconjugated, unconjugated bilirubin is reabsorbed leading to entero-hepatic circulation, which plays a significant role in the development on neonatal jaundice.

Previous studies have shown that early meconium evacuation was associated with lower total serum bilirubin levels and decreased risk for clinically significant neonatal jaundice (Jirsova, DeCarvalho, Boyer, Gourley, Salariya and Gourley). Other studies in healthy term neonates have shown no benefit from rectal glycerin in reducing peak serum bilirubin levels. Bader et al performed a prospective study to evaluate the general effect of glycerin suppository administration in reducing total serum bilirubin levels in healthy term neonates. Glycerin suppositories were given immediately after birth and every 4 hours thereafter, until evacuation of first stool. The suppositories had no effect on mean total serum bilirubin levels at 48 hours of age. It was concluded that glycerin suppositories should not be routinely recommended as a means for reducing the severity of neonatal jaundice. However, it was found that in a subgroup of male infants with blood group type A there were significantly lower mean total serum bilirubin levels after induction of earlier meconium evacuation with glycerin suppositories. Weisman et al performed a similar prospective study in healthy term neonates and found that giving glycerin suppositories does hasten the passage of meconium and transitional stool; however, there was no effect on peak serum bilirubin levels during the first 3 days of life and no effect on need for phototherapy. Chen et al described a prospective, randomized controlled trial with two groups of healthy term neonates. The experimental group received glycerin enemas at 30 minutes and 12 hours of life. Bilirubin levels were followed for the first 7 days of life. The intervention had no effect on peak serum bilirubin levels or serum bilirubin levels in the first 7 days of life.

No data exist on the use of glycerin suppositories in premature neonates, although its use is a common practice to increase meconium clearance and stooling in the case of hyperbilirubinemia. However, it may not be a justified practice, based on data for full-term infants. Experts argue that premature neonates may have upward of 25% more enterohepatic circulation than full-term neonates (S. Amin, personal communication). Therefore, because premature neonates have the potential to recirculate bilirubin, increasing stool frequency through schedule glycerin suppositories might play a therapeutic role in the management of hyperbilirubinemia in this population.

It is a common practice in our unit to provide glycerin suppositories every 8 hours to infants under phototherapy in an attempt to more rapidly reduce bilirubin levels by decreasing enterohepatic circulation of unconjugated bilirubin. This practice is not evidence-based, nor is it standard practice in many NICUs throughout the country. Glycerin suppositories are not without risk. They can lead to rectal fissures and tears, bloody stools and unnecessary vagal stimulation.

If administration of glycerin shaves decreases length of phototherapy to a clinically significant extent, there may be improved success with feedings including breastfeeding, improved infant-parent bonding, shortened length of stay and overall increased family satisfaction. However, if glycerin suppositories are not shown to reduce duration of phototherapy, reduce peak total serum bilirubin (TSB) levels, reduce the number of TSB levels drawn and increase the rate of decline of hyperbilirubinemia, then a potentially useless therapy with potential for untoward side effects may be avoided.

ELIGIBILITY:
Inclusion Criteria:

1. Baby born between 30 to 34 6/7 weeks gestational age (GA) at birth and admitted to NICU
2. Baby with physiologic hyperbilirubinemia requiring phototherapy by current NICU criteria.
3. Parental permission.

Exclusion Criteria:

1. Babies less than 30 weeks GA or greater than 34 6/7 weeks GA
2. Non-physiologic hyperbilirubinemia: (1) positive Coombs test and (2) hematocrit < 5th percentile for GA (see Jopling J, Henry E, Wiedmeier SE, Christensen RD, Reference. Ranges for Hematocrit and Blood Hemoglobin Concentration During the Neonatal Period: Data From a Multihospital Health Care System. Pediatrics 2009; 123(2):e333 -e337.) and (3) ABO or Rh incompatibility.
3. Any infant with bilirubin level within 2 mg/dL of exchange transfusion.
4. Any infant who has phototherapy started prior to reaching light level (prophylactic)
5. Baby with any GI abnormalities such as NEC, intestinal perforation, gastroschisis, omphalocele, malrotation and or volvulus, duodenal atresia, intestinal strictures/adhesions, imperforate anus.
6. Any infant begun on triple or greater phototherapy at time of initiation of treatment.
7. Any infant judged by the attending physician to be placed at increased risk by study participation.

Ages: 30 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2012-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meggan Butler-O'Hara, RN, MSN, PNP, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center NICU, Rochester, New York, United States

REFERENCES:
- [Background] Maisels MJ. Jaundice. In: Avery GB, Fletcher MA, MacDonald MG, eds. Neonatology: Pathophysiology and Management of the Newborn. Philadelphia: Lippincott Williams and Wilkins; 1999:765-819.
- [Background] Rosta J, Makoi Z, Kertesz A. Delayed meconium passage and hyperbilirubinaemia. Lancet. 1968 Nov 23;2(7578):1138. doi: 10.1016/s0140-6736(68)91603-6. No abstract available. PMID 4177180
- [Background] Porto SO. Jaundice in congenital malrotation of the intestine. Am J Dis Child. 1969 Jun;117(6):684-8. doi: 10.1001/archpedi.1969.02100030686011. No abstract available. PMID 5771508
- [Background] Jirsova V, Janovsky M. Hyperbilirubinemia connected with parenteral administration of higher amounts of fluids in premature infants. Biol Neonate. 1978;33(3-4):132-4. doi: 10.1159/000241062. PMID 98182
- [Background] De Carvalho M, Robertson S, Klaus M. Fecal bilirubin excretion and serum bilirubin concentrations in breast-fed and bottle-fed infants. J Pediatr. 1985 Nov;107(5):786-90. doi: 10.1016/s0022-3476(85)80418-2. PMID 4056981
- [Background] Boyer DB, Vidyasagar D. Serum indirect bilirubin levels and meconium passage in early fed normal newborns. Nurs Res. 1987 May-Jun;36(3):174-8. PMID 3646618
- [Background] Bader D, Yanir Y, Kugelman A, Wilhelm-Kafil M, Riskin A. Induction of early meconium evacuation: is it effective in reducing the level of neonatal hyperbilirubinemia? Am J Perinatol. 2005 Aug;22(6):329-33. doi: 10.1055/s-2005-871529. PMID 16118723
- [Background] Weisman LE, Merenstein GB, Digirol M, Collins J, Frank G, Hudgins C. The effect of early meconium evacuation on early-onset hyperbilirubinemia. Am J Dis Child. 1983 Jul;137(7):666-8. doi: 10.1001/archpedi.1983.02140330050013. PMID 6858980
- [Background] Chen JY, Ling UP, Chen JH. Early meconium evacuation: effect on neonatal hyperbilirubinemia. Am J Perinatol. 1995 Jul;12(4):232-4. doi: 10.1055/s-2007-994460. PMID 7575822
- [Background] Amin, S. (2011). Personal communication.
- [Background] Jopling J, Henry E, Wiedmeier SE, Christensen RD. Reference ranges for hematocrit and blood hemoglobin concentration during the neonatal period: data from a multihospital health care system. Pediatrics. 2009 Feb;123(2):e333-7. doi: 10.1542/peds.2008-2654. PMID 19171584

RESULTS

PARTICIPANT FLOW:
Groups:
- Glycerin Suppository: Based on our institution's protocol, infant will receive a glycerin shave within one hour of initiation of phototherapy and then every eight hours while under phototherapy.
  Subjects will be block randomized (varying block sizes of 2 to 8). Babies in both groups will be fed according to NICU standard birth weight protocols. Stratified enrollment will occur with 2 separate groups:
  1. Infants who are NPO (< 20 mL/kg/day of fluids enterally at the time of therapy) vs.
  2. Those being enterally fed at least 20 mL/kg/day of total fluids at the time of therapy.
  Phototherapy: Light therapy is used to treat cases of neonatal jaundice through the isomerization of the bilirubin and consequently transformation into compounds that the newborn can excrete via urine and stools.
  glycerin suppository: Promotes stooling through rectal stimulation and softening of stool. Given every 8 hours rectally. A pediatric glycerin suppository is 1.2 grams.
- No Glycerin Suppository: Infants will receive no scheduled glycerin suppositories, while under phototherapy (unless otherwise directed by attending physician).
  Subjects will be block randomized (varying block sizes of 2 to 8). Babies in both groups will be fed according to NICU standard birth weight protocols. Stratified enrollment will occur with 2 separate groups:
  1. Infants who are NPO (< 20 mL/kg/day of fluids enterally at the time of therapy) vs.
  2. Those being enterally fed at least 20 mL/kg/day of total fluids at the time of therapy.
  Phototherapy: Light therapy is used to treat cases of neonatal jaundice through the isomerization of the bilirubin and consequently transformation into compounds that the newborn can excrete via urine and stools.
Period: Overall Study
Arm/Group | Glycerin Suppository | No Glycerin Suppository
Started | 40 | 39
Completed | 40 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Demographic data, including age at start of phototherapy, was incomplete, missing for one infant in each study group.
Groups:
- Glycerin Suppository: Based on our institution's protocol, infant will receive a glycerin shave within one hour of initiation of phototherapy and then every eight hours while under phototherapy.
  Subjects will be block randomized (varying block sizes of 2 to 8). Babies in both groups will be fed according to NICU standard birth weight protocols. Stratified enrollment will occur with 2 separate groups:
  1. Infants who are NPO (< 20 mL/kg/day of fluids enterally at the time of therapy) vs.
  2. Those being enterally fed at least 20 mL/kg/day of total fluids at the time of therapy.
  Phototherapy: Light therapy is used to treat cases of neonatal jaundice through the isomerization of the bilirubin and consequently transformation into compounds that the newborn can excrete via urine and stools.
  glycerin suppository: Promotes stooling through rectal stimulation and softening of stool. Given every 8 hours rectally. A pediatric glycerin suppository is 1.2 grams. All infants in this study arm will receive our
- Total: Total of all reporting groups
Arm/Group | Glycerin Suppository | No Glycerin Suppository | Total
Number analyzed (Participants) | 39 | 38 | 77
Age, Continuous [Mean (Standard Deviation); unit: hours] | 62.2 (19.1) | 72.7 (25.2) | 67.4 (22.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 19 | 18 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 8 | 15
  White | 31 | 26 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 39 | 38 | 77
Birth Weight [Mean (Standard Deviation); unit: grams] — All participants that started the study were included in this baseline measure description.
  grams | 1792 (513) | 1933 (315) | 1862 (415)
First observed total bilirubin [Mean (Standard Deviation); unit: mg/dL] — All participants that started the study were included in this baseline measure description.
  mg/dL | 8.1 (3.0) | 8.3 (3.3) | 8.2 (3.1)
Gestation age [Mean (Standard Deviation); unit: weeks] — All participants that started the study were included in this baseline measure description.
  weeks | 33.2 (1.4) | 33.0 (1.1) | 33.1 (1.3)
Feeding stratum [Number; unit: participants] — NPO is infants receiving ≤ 20 mL/kg/day of fluids enterally at the time of therapy PO is infants being enterally fed > 20 mL/kg/day of total fluids at the time of therapy.
  All participants that started the study were included in this baseline measure description.
  participants
    NPO | 18 | 16 | 34
    PO-formula | 7 | 7 | 14
    PO -breastmilk | 7 | 6 | 13
    PO-both formula and breastmilk | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Hours of Required Phototherapy
Time Frame: from time of enrollment to time of discharge, for a maximum of 10 weeks
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Glycerin Suppository | No Glycerin Suppository
Number analyzed (Participants) | 40 | 39
hours | 72 (49) | 61 (53)

2. Secondary Outcome: Number of Episodes of Repeat Phototherapy
Description: Bilirubin levels are checked at regular intervals after phototherapy is discontinued to make sure levels are safe. Depending on rate of rise and predetermined "unsafe" bilirubin level, phototherapy may be restarted.
Time Frame: from time of enrollment to time of discharge, for a maximum of 10 weeks
Measure: Median (Full Range); unit: episodes of repeat phototherapy
Arm/Group | Glycerin Suppository | No Glycerin Suppository
Number analyzed (Participants) | 40 | 39
episodes of repeat phototherapy | 0 [0 to 7] | 0 [0 to 7]

3. Secondary Outcome: Peak Total Serum Bilirubin Level
Description: Bilirubin levels were checked every 12 hours while the infant was under phototherapy. A bilirubin level was then to be checked at least twice, 8-12 hours or longer apart, following discontinuation of phototherapy.
Time Frame: from time of enrollment to time of discharge every 12 hours while under phototherapy, for a maximum of 10 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Glycerin Suppository | No Glycerin Suppository
Number analyzed (Participants) | 40 | 39
mg/dL | 11.3 (1.8) | 12.0 (1.5)

4. Secondary Outcome: Rate of Decline in Bilirubin Levels (mg/dL/hr)
Description: Absolute change over time from peak to first discontinuation of phototherapy lights
Time Frame: from time of enrollment to time of discharge, for a maximum of 10 weeks
Measure: Mean (Standard Deviation); unit: mg/dL/hr
Arm/Group | Glycerin Suppository | No Glycerin Suppository
Number analyzed (Participants) | 40 | 39
mg/dL/hr | 0.4 (0.2) | 0.4 (0.1)

5. Secondary Outcome: Length of Initial Round of Phototherapy
Description: time start to time finally off phototherapy, including any breaks during which they were off
Time Frame: from time of enrollment to time of discharge, for a maximum of 10 weeks
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Glycerin Suppository | No Glycerin Suppository
Number analyzed (Participants) | 40 | 39
hours | 118 (128) | 81 (85)

ADVERSE EVENTS:
Arm/Group | Glycerin Suppository | No Glycerin Suppository
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 1/40 | 0/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glycerin Suppository (N=40) | No Glycerin Suppository (N=39)
Bloody Stool (Gastrointestinal disorders) | 1 (1) | 0 (0) — One infant in the glycerin suppository group had blood streaks in the stool, but this was after a non-indicated glycerin shave, given in error following the discontinuation of phototherapy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes